CLINICAL TRIAL: NCT03983486
Title: Use of Imaging Flow Cytometry for Immunophenotyping Coupled With Cytogenetic Abnormalities Detection by Fluorescent in Situ Hybridization (FISH) and Applicability in Cytogenetic Risk Stratification of Multiple Myeloma (CIF-PM)
Brief Title: Rationale for Cytogenetic Risk Stratification by Imaging Flow Cytometry in Multiple Myeloma
Acronym: CIF-PM
Status: Withdrawn | Type: Observational
Why Stopped: technical problem
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0002
Record Dates: First submitted 2018-04-13; First posted 2019-06-12 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma
Keywords: IS-FISH; Imaging flow cytometry; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Imaging flow cytometry in multiple myeloma — Combination of immunophenotyping by flow cytometry and FISH in suspension (IS-FISH) may provide both cytogenetic and phenotypic information for a large number of cells in a single test. In this scope, a recent study demonstrated a proof of concept for IS-FISH to detect non pathological signals with the new ImageStream X technology (ISX).1

SUMMARY:
A pioneer study demonstrated a proof of concept for IS-FISH with the new ISX technology. This state of the art technology has been recently acquired by the CHU of Amiens. In the present study the investigators want to establish a workflow for simultaneous immunostaining and characterization of FISH cytogenetic pathological signals with the imaging flow cytometer ISX, such as chromosomic gains, losses and translocations in multiple myeloma (MM). The gold standard technology for the detection of prognostic cytogenetic aberrations in MM is a FISH analysis after bone marrow (BM) plasma cells sorting (PCS).2,3 In MM, plasma cells isolation is usually based on CD38 and/or CD138 expression. Cytogenetic risk stratification is guided by the detection of 4 chromosomal aberrations: TP53 and CDKN2C deletions, CKS1B gains and t(4;14) translocation. Thanks to ISX technology the investigators may avoid cumbersome task of cell sorting (outsourced service for our hospital) meanwhile measuring precisely and qualitatively aberrant FISH signals on a large amount of cells.

DETAILED DESCRIPTION:
In a first time (period of 6 months), the development will be performed on CD38 and/or CD138 expressing cell lines. Regular FISH protocols will be finely tuned to fit immunophenotyping and cells in suspension constraints needed in IS-FISH. In a second time, the protocol will be applied to MM BM. Cells from BM aspiration will be processed and analysed on the ISX in Amiens. Based on last years local activity, this step is expected to last 2 years, so as to be able to obtain 5 samples from patients harbouring of each prototypical cytogenetic aberration above described. Inclusions will be guided by the results of PCS conducted before the first treatment initiation. Finally the results will be compared with PCS.

ELIGIBILITY:
Inclusion Criteria:

* Available BM samples from active MM patients followed in the CHU of Amiens will be selected on the basis of PCS analysis systematically performed before treatment initiation.
* signed consent

Exclusion Criteria:

* <5% plasma cells in BM.
* Pre-bone marrow autograft samples

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with multiple myeloma (MM)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Detection of plasmocytes by imaging flow cytometry techniques in plasmocytes cell line. | during the first six months of the study
  In a first time (period of 6 months), the development will be performed on CD38 and/or CD138 expressing cell lines. Regular FISH protocols will be finely tuned to fit immunophenotyping and cells in suspension constraints needed in IS-FISH (FISH in suspension).
  Development of the technique of the first period will be made in order to test :
  * the ability to measure FISH and immunostaining signals simultaneously
  * the ability to count a number of FISH spots consistent with ploidy (eg 1 X centromeric signal for men, 2 for women).
Detection of plasmocytes by imaging flow cytometry techniques in multiple myeloma bone marrow (MM BM). | from 6 months after the beginning of the study to two years after the beginning of the study
  Cells from BM (bone marrow) aspiration will be processed and analyzed on the ISX (Image Stream X technology) in Amiens.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No